CLINICAL TRIAL: NCT07025824
Title: Randomized Evaluation of Treosulfan Versus Melphalan Conditioning Followed by PTCy in Patients With AML and MDS Undergoing Allogeneic Transplantation
Brief Title: Evaluation of Treosulfan Versus Melphalan Conditioning Followed by PTCy in Patients With AML and MDS Undergoing Allogeneic Transplantation
Acronym: RELEVANT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: medac GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TUD-ETAL-5-084
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: AML - Acute Myeloid Leukemia; MDS (Myelodysplastic Syndrome)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts | interventions — treosulfan; Melphalan; Honey; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treo - Arm (Experimental): Treo d-4 - d-2 + Flud d-6 till d-2
  Interventions: Drug: Treosulfan (Treo); Drug: Fludarabine (Flud)
- MEL - Arm (Active Comparator): Mel d-2 + Flud d-6 till d-2
  Interventions: Drug: Melphalan (Mel); Drug: Fludarabine (Flud)

INTERVENTIONS:
Drug: Treosulfan (Treo) — 10 g/m2 intravenous
  Arms: Treo - Arm
Drug: Melphalan (Mel) — 140 mg/m2 intravenous
  Arms: MEL - Arm
Drug: Fludarabine (Flud) — 30 mg/m2 intravenous

SUMMARY:
The aim of this study is to compare the effectiveness and tolerability of two conditioning chemotherapies prior to allogeneic stem cell transplantation.

The following will also be investigated:

* Survival
* Remission and Relapse rate
* Engraftment or graft failure
* Graft versus Host Disease (GvHD)

ELIGIBILITY:
Main Inclusion Criteria:

1. Informed consent signed by the patient capable of giving
2. Patient scheduled for allogeneic transplantation within the next 3 weeks
3. Age ≥ 18 years
4. AML or MDS according to WHO with indication for allogeneic HCT:

   1. AML in first or second complete remission (CR) or complete remission with incomplete hematologic recovery (CRi/CRh) or morphologic leukemia-free state (MLFS)
   2. MDS according to WHO
5. Increased risk for treatment-related toxicity by myeloablative conditioning according to at least one of the following criteria:

   1. Patients aged ≥ 50 years at transplant and/or
   2. HCT-CI > 2 and/or
   3. AML or MDS scheduled for 2nd allogeneic HCT from different donor with minimum of 12 months after 1st allogeneic HCT
6. Availability of a suitable donor:

   1. Matched sibling donor (MSD) or
   2. matched unrelated donor (MUD, 10/10 HLA) or
   3. mismatched unrelated donor (MMUD, single allele or antigen mismatch at HLA-A, -B, -C, or -DRB1 and no concurrent -DQB1 mismatch (9/10) shown by confirmatory typing) or
   4. haploidentical family donor
7. Planned GvHD prophylaxis with standard PTCy (with 50mg/kg body weight on days +3 and +4)
8. No history of cardiac disease that preclude allogeneic HCT and absence of active symptoms, otherwise, documented left ventricular ejection fraction

   * 40 %.
9. No need for supplementary oxygen on day of randomization

Main Exclusion Criteria:

1. Patients with acute promyelocytic leukemia with t(15;17)(q22;q12)
2. Patients with graft failure after previous allogeneic HCT
3. Patients with scheduled 2nd allogeneic HCT within 12 months after 1st allogeneic HCT
4. Pretreatment with either melphalan or treosulfan within the last 12 months prior to randomization
5. Planned TBI as part of conditioning
6. Severe organ dysfunction defined by either one of the following criteria:

   1. Serum bilirubin > 1.5 × ULN (if not considered Gilbert-syndrome) or
   2. ALAT or ASAT > 5 × ULN
7. Uncontrolled infection at the time of randomization.
8. Active viral hepatitis unless serology demonstrates clearance of infection. Occult or prior hepatitis B virus (HBV) infection, defined as negative hepatitis B surface antigen and positive total hepatitis core antibodies, may be included if HBV DNA is undetectable, provided that patients are willing to undergo monthly DNA testing. Patients who have protective titers of hepatitis B surface antibody after vaccination or prior cured hepatitis B are eligible. Patients for hepatitis C virus (HCV) antibody are eligible provided PCR if negative for HCV RNA.
9. Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
overall survival (OS) | 2 years after randomization

SECONDARY OUTCOMES:
non-relapsed mortality (NRM) | 2 years after randomization
relapse-free survival (RFS) | 2 years after randomization
-Cumulative incidences of acute and chronic GvHD | 2 years after randomization
Rates of AEs/SAEs/AESI | 56 days after allogeneic stem cell transplantation
-Cumulative incidence of relapse (CIR) | 2 years after randomization
-Rate of engraftment on day +28 | 2 years after randomization
Rate of morphologic and molecular CR/CRh/CRi/MLFS | day +56 after allogeneic stem cell transplantation

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (4):
  - Medizinische Fakultät der TU Dresden, Medizinische Klinik und Poliklinik I, Dresden
  - Universitätsmedizin Halle (Saale), Halle
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Universitätsklinikum Münster, Medizinische Klinik A, KMT-Zentrum, Münster